CLINICAL TRIAL: NCT02297724
Title: MRI Assessment of Placental Health
Status: Recruiting | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); Massachusetts Institute of Technology (Other); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH); Madrid-MIT M+Visión Consortium (Unknown)
Responsible Party: Principal Investigator, Ellen Grant, Director, Fetal-Neonatal Neuroimaging and Developmental Science Center, Boston Children's Hospital
Other Study IDs: CHB_Placenta2013; R01EB017337-01 (NIH)
Record Dates: First submitted 2014-10-15; First posted 2014-11-21 (Estimated); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Intrauterine Growth Restriction
MeSH Terms: conditions — Fetal Growth Retardation | interventions — Oxygen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- all subjects: For all subjects, administration of oxygen will last for no more than 10 min, with flow rate 15L/min via non-rebreather facial mask. Each subject will have once of the administration per scan. Data collection will start about 10 min before the administration of oxygen, and last throughout the oxygen exposure, then continue for about 10 min after oxygen exposure for each subject.
  Interventions: Other: Oxygen

INTERVENTIONS:
Other: Oxygen — Administration of oxygen will last for no more than 10 min, with flow rate 15L/min via non-rebreather facial mask. Each subject will have once of the administration per scan.

SUMMARY:
The ultimate goal of this project is to develop methods that allow informed decision-making on the delivery time of fetuses that are at increased risk of stillbirth due to IUGR. In placenta related IUGR pregnancies, there can be multiple concurrent placental pathologies. Although there is no specific correspondence between a single type of pathology and IUGR, the common result of these pathologies is placental insufficiency, which limits the maternal-fetal exchange. Oxygen and nutrition transport is known to be hindered in IUGR placentas due to obstructed or abrupt vasculature, massive fibrin deposition, and inflammation in the villous and intervillous space (villitis). Thus one potential approach to distinguish IUGR pregnancies from normal ones is to assess the efficiency of placental transport. Based on the hypothesis that efficiency of oxygen transport is representative for overall oxygen and nutrition transport in placenta, the investigators propose to characterize the blood oxygenation and blood perfusion in placenta in vivo via MRI, and use it as an index for better stratification in the IUGR risk group. The investigators will also consider alternative MRI approaches such as structural, diffusion and spectroscopy measurements inside the placenta, which might reflect the state of placental transport and reveal the status of placental health.

Specific aims: 1) To correlate the MRI metrics that differentiate placental insufficiency from normal placenta transport with histopathology data of the placenta. 2) To correlate the MRI metrics that reflects placental insufficiency with fetal outcome

ELIGIBILITY:
Inclusion Criteria:

1. The pregnant mother with twin gestation with diagnosis of selective IUGR based upon obstetrical US findings as following:

   * Proven monochorionicity / dichorionicity
   * Discordance in estimated fetal weight (EFW). Growth restriction (<10 percentile of norm) in one or both fetus(es) AND/OR growth discordance (> or = 20%) between twin fetuses.
2. The pregnant mother with singleton gestation with diagnosis of IUGR based upon obstetrical US findings as following:

   * Proven singleton gestation
   * Growth restriction of fetus (<10 percentile of norm)
   * Doppler measurements that indicates placental insufficiency: umbilical artery, middle cerebral artery, uterine artery; or oligohydramnios.
3. Gestational age: Bigger than 18 weeks.
4. Pregnant mother is between age 18 to 45, clinically stable and can safely tolerate fetal MRI study.

Exclusion Criteria:

Fetuses/infants with the following features will be excluded.

1. Fetus/infant with chromosomal anomalies or known genetic disorders.
2. Fetus/infant with other major congenital malformation.
3. Presence of any condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient, quality or completeness of the data.

Pregnant mothers with the following features will be excluded.

1. Mothers with contraindication to MRI (with pacemaker, metal in body, oversize).
2. Mothers with claustrophobia
3. Mothers medically unstable for the MRI study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * pregnant mothers with twin gestation with diagnosis of selective IUGR
  * pregnant mothers with singleton gestation with diagnosis of IUGR
  * singleton pregnant mothers and twin pregnant mothers with no apparent medical complication on fetuses
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2014-04; Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
BOLD MRI signal change during maternal oxygen exposure in placenta and fetus | 30 min during the 1 hour scan
placental volume on MRI image | 5 min during 1 hour scan

SECONDARY OUTCOMES:
pathological reports of placenta after delivery | 1 day
fetal growth curve after birth | up to 6 month

CONTACTS AND LOCATIONS:
Overall Officials: Patricia E Grant, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- Boston Children's Hospital, Boston, Massachusetts, United States
- Hospital Universitario de Fuenlabrada, Madrid, Spain